CLINICAL TRIAL: NCT00580970
Title: A Phase II Study to Prevent Radiation-Induced Rectal Injury With Lovastatin
Brief Title: Study of Effectiveness of Lovastatin to Prevent Radiation-Induced Rectal Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-10802; NCI-2011-01676 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radiation therapy; lovastatin; rectal injury
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lovastatin for 1 yr (Experimental): Lovastatin (20-80 mg/d) was started on day 1 of radiation and continued for 12 months. Patients were followed for an additional 12 months. Lovastatin once per day for 1 year. After the implant, they are asked to return for checkups (study visits 4-13) 4 weeks, 8 weeks, 4 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months and 24 months after the procedure. At 8 weeks, 4 months, 6 months, 9 months and 12 months, will also have a blood test to check their liver.
  Interventions: Drug: lovastatin

INTERVENTIONS:
Drug: lovastatin — The HMG-coA reductase inhibitor used in this study will be lovastatin. Dosage: 20 mg/d PO with evening meal. Patients on a higher dose of lovastatin at the time of study entry may continue at that dose level; for patients switching to lovastatin, the dose will be at the discretion of the prescribing physician, but must be at least 20 mg/day.Schedule: begin on the first day of external beam radiation therapy (external beam alone or external beam followed by brachytherapy) or on the day of brachytherapy (brachytherapy alone or brachytherapy followed by external beam radiotherapy) and continue for 12 months. Patients or their third party payers will be expected to cover the cost of the drug.
  Other Names: Altoprev; Mevacor

SUMMARY:
Lovastatin may protect against late effects of radiation therapy in patients with prostate cancer

DETAILED DESCRIPTION:
Oral lovastatin will be given at the dose of 20 mg/day with evening meal beginning on the first day of external beam radiation therapy (external beam alone or external beam followed by brachytherapy) or on the first day of brachytherapy (brachytherapy alone or brachytherapy followed by external beam radiotherapy) and continue for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate
* Planned treatment with radiation therapy to include external beam and/or brachytherapy with curative intent (total dose ≥60 Gy). A portion of the rectum must receive at least 60 Gy.
* Age at least 18 years
* Karnofsky Performance Status (KPS) ≥ 70
* No history of prior radiotherapy to the prostate or rectum
* History of prior malignancy, if likely to live at least 4 years, is acceptable.
* No evidence of distant metastases
* Patients may be taking an HMG-coA-reductase inhibitor, but to be eligible, they must be able to be changed to lovastatin 20 mg/day, with the permission of their prescribing physician.
* Creatine kinase < 5 times upper normal limit
* Sufficient renal function defined as calculated creatinine clearance ≥ 30ml/min
* transaminases < 3 times upper normal limit

Exclusion Criteria:

* Planned abdomino-perineal resection after radiotherapy
* Contraindication to an HMG-coA-reductase inhibitor
* Major medical or psychiatric illness, which in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.
* Currently taking an inhibitor of cytochrome P450 3A4
* Active liver or muscle disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S. Anscher, MD, Principal Investigator — Massey Cancer Center
Locations (3):
- United States (3):
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Massey Cancer Center/Virginia Commonwealth University, Richmond, Virginia
  - Southside Regional Medical Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was between between 2007 to 2013 at Virginia Commonwealth University, Stony Point, Hanover Medical Center, Southside Regional Medical Center, and Hunter Holmes McGuire Veterans Affairs Medical Center (VAMC).
Pre-assignment Details: Enrollment period was between April 12, 2007 and May 30, 2013. During that time 73 consecutive subjects enrolled in the study, 72 started treatment. A total of 20 subjects were ineligible for analysis because they did not reach 6 months of Lovastatin treatment, resulting in a total of 53 evaluable subjects.
Groups:
- Supportive Care (Lovastatin): Subjects took Lovastatin on the first day of radiation (either EBRT,external beam radiotherapy, or on the day of brachytherapy) and continued for 12 months.
  73 subjects enrolled in the study, 72 started treatment, 20 subjects were ineligible for analysis, and a total of 53 evaluable subjects.
Period: Pre-treatment
Arm/Group | Supportive Care (Lovastatin)
Started | 73
Completed | 72
Not Completed | 1
Not completed — Non-compliance | 1
Period: Treatment (Lovastatin)
Arm/Group | Supportive Care (Lovastatin)
Started | 72
6 Months of Treatment | 53 (Subjects evaluable for analysis)
Completed | 53
Not Completed | 19
Not completed — Non-compliance | 6
Not completed — Intolerance of Lovastatin | 7
Not completed — Physician Decision | 4
Not completed — Development of metastatic second primary | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Between April 12, 2007 and May 30, 2013, 73 consecutive patients enrolled in the study. A total of 20 patients did not complete at least 6 months of Lovastatin treatment and were deemed ineligible for the purpose of assessing late rectal toxicity and additional patients were enrolled in order to achieve the accrual goal of 53 evaluable patients.
Groups:
- Supportive Care (Lovastatin) (Evaluable): The 53 subjects started Lovastatin treatment on the first day of radiation (either EBRT,external beam radiotherapy, or on the day of brachytherapy) and continued up to 12 months. The subjects were considered evaluable for analysis because they completed 6 months of Lovastatin.
- Supportive Care (Lovastatin) (Ineligible): The 20 subjects started Lovastatin on the first day of radiation (either EBRT,external beam radiotherapy, or on the day of brachytherapy). The subjects were ineligible because they did not complete 6 months of Lovastatin.
- Total: Total of all reporting groups
Arm/Group | Supportive Care (Lovastatin) (Evaluable) | Supportive Care (Lovastatin) (Ineligible) | Total
Number analyzed (Participants) | 53 | 20 | 73
Age, Continuous [Median (Full Range); unit: years] | 63 [47 to 80] | 58.5 [50 to 69] | 62 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 53 | 20 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 10 | 32
  White | 31 | 10 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 20 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Physician Reported Rectal Toxicity ≥ Grade 2 During the First 2 Years of Radiation Treatment
Description: The primary endpoint of this study was percentage of participants with physician reported rectal toxicity ≥Grade 2 during the first 2 years after treatment. A one sided test will be conducted in order to evaluate reduction of risk from adding Lovastatin. The analysis is using a one-stage design, 5% level of significance, and 83% power.
Time Frame: 24 months
Population: The primary endpoint of the study was percentage of participants with physician reported rectal toxicity ≥Grade 2 during the first 2 years after treatment. Only the highest-grade toxicity for each symptom was counted. Symptoms starting in the acute period and unresolved beyond 90 days post treatment are considered late toxicity.
Measure: Number; unit: percentage of participants
Arm/Group | Supportive Care (Lovastatin) (Evaluable)
Number analyzed (Participants) | 53
percentage of participants | 38
Statistical Analysis 1: Comparison: Supportive Care (Lovastatin) (Evaluable); Test type: Superiority or Other; p = 0.9138, t-test, 1 sided — Considering all late rectal toxicities, 38% (20/53) of participants developed physician reported Grade 2 or higher GI toxicity during 2 year follow up. The threshold for significance was p < 0.05; A one sided t-test, with 5% level of significance, and 83% power was used which required 53 subjects

ADVERSE EVENTS:
Time Frame: 2 years
Description: Systematic Assessments includes medical history, physical exam, Karnofsky Performance Status (KPS), International Index of Erectile Function (IIEF), The Expanded Prostate Cancer Index Composite (EPIC), Common Terminology Criteria for Adverse Events Version 3 (CTCAE), and blood samples (e.g. Lipid profile, CK, CPC, Hepatic panel).
Groups:
- Supportive Care (Lovastatin): Subjects who started treatment on Lovastatin on the first day of radiation therapy (external beam radiation therapy (EBRT) alone, brachytherapy alone, or EBRT followed by brachytherapy).
  73 subjects enrolled in the study, 72 started Lovastatin treatment, 20 subjects were ineligible for analysis, and a total of 53 subjects evaluable for analysis. 72 subjects started treatment and were at risk for Adverse Events (AEs) and Serious Adverse Events(SAEs).
Arm/Group | Supportive Care (Lovastatin)
Serious Adverse Events (participants affected / at risk) | 8/72
Other Adverse Events (participants affected / at risk) | 70/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Lovastatin) (N=72)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) — Blood/Bone Marrow
Cardiac General (Cardiac disorders) | 1 (1)
Gastrointestinal/Proctitis (Gastrointestinal disorders) | 1 (1)
Hemorrhage/Bleeding (Gastrointestinal disorders) | 1 (1) — Colon
Hemorrhage/Bleeding (Gastrointestinal disorders) | 1 (1) — Lower GI NOS
Hemorrhage/Bleeding (Gastrointestinal disorders) | 1 (2) — GI - Rectum
Hepatobiliary/Pancreas (Gastrointestinal disorders) | 1 (1) — Pancreatitis
Pain (General disorders) | 1 (1) — Chest/thorax Not Otherwise Specified (NOS)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Lovastatin) (N=72)
Hot flashes/flushes (Endocrine disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 12 (21)
Diarrhea (Gastrointestinal disorders) | 48 (94)
Flatulence (Gastrointestinal disorders) | 48 (108)
Hemorrhage, GI - Anus (Gastrointestinal disorders) | 17 (29)
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 5 (6)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 9 (15)
Hemorrhoids (Gastrointestinal disorders) | 6 (8)
Incontinence, anal (Gastrointestinal disorders) | 19 (34)
Nausea (Gastrointestinal disorders) | 4 (5)
Pain - Abdomen NOS (Gastrointestinal disorders) | 10 (13)
Proctitis (Gastrointestinal disorders) | 25 (35)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 (9)
Pain - Back (Musculoskeletal and connective tissue disorders) | 6 (10)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 6 (10)
Bladder spasms (Renal and urinary disorders) | 26 (50)
Cystitis (Renal and urinary disorders) | 41 (64)
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 15 (22)
Incontinence, urinary (Renal and urinary disorders) | 33 (75)
Dysuria (Renal and urinary disorders) | 12 (14)
Stricture/stenosis (including anastomotic), GU - Prostate (Renal and urinary disorders) | 6 (13)
Urinary frequency/urgency (Renal and urinary disorders) | 52 (108)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 21 (36)
Erectile dysfunction (Reproductive system and breast disorders) | 8 (8)
Pain - Penis (Reproductive system and breast disorders) | 4 (5)
Pain - Urethra (Reproductive system and breast disorders) | 7 (11)
Nocturia (Renal and urinary disorders) | 5 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No